CLINICAL TRIAL: NCT00141739
Title: The Addition of Etanercept to Standard GVHD Prophylaxis in Patients Undergoing a Full Intensity Allogeneic Hematopoietic Stem Cell Transplant for the Prevention of Transplant Related Complications
Brief Title: Study of Etanercept for the Prevention of Complications Resulting From Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004.008
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Graft-Versus-Host Disease
Keywords: Stem Cell Transplantation; Graft-Versus-Host Disease; prophylaxis
MeSH Terms: conditions — Graft vs Host Disease | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GVHD prophylaxis (Experimental): GVHD prophylaxis with etanercept
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 0.4 mg/kg per dose [maximum dose 25 mg] SC for prophylaxis. To start in the 24 hour time period along with the initiation of the preparative regimen for the stem cell transplant.
  Etanercept will be administered twice weekly until day +56 (8 weeks) post transplant.
  Other Names: Enbrel

SUMMARY:
This is a clinical trial to see if the addition of etanercept to standard preventative medicines helps in preventing two major complications of hematopoietic stem cell transplantation (HSCT): decrease the rate of acute graft-vs-host disease (GVHD) and the risk of death.

DETAILED DESCRIPTION:
This is a clinical trial to see if the addition of etanercept helps in preventing two major complications of hematopoietic stem cell transplantation (HSCT). The main objective will be to see whether the addition of etanercept to standard preventative medicines will decrease the rate of acute graft-vs-host disease (GVHD) and the risk of death by 100 days following allogeneic HSCT from volunteer donors.

GVHD is a common complication following a bone marrow transplant from another donor. GVHD occurs after transplant when the donor's blood cells recognize parts of the body as foreign. During this process, chemicals called cytokines are released that may damage certain body tissues, including the gut, liver and skin. Some of the main effects can include red skin rash, diarrhea, sometimes with blood, and yellow jaundice. It can range from mild to life threatening and often requires admission to the hospital for treatment. The standard treatment for acute GVHD is a combination of steroids and another drug that suppress the immune system, such as tacrolimus or cyclosporine.

Etanercept is a drug that blocks a chemical called Tumor Necrosis Factor (TNF) from causing damage to your tissue. The purpose of etanercept is to help improve the response to standard treatment for GVHD. Previous studies have shown that less than 50% of patients respond fully to GVHD treatment. Without a good response, patients often have a prolonged treatment for this disease, often involving hospitalization and sometimes even death. Etanercept (Enbrel) will be added to the standard treatment to see if we can lower the rate of GVHD and the risk of death from GVHD by blocking TNF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 1 and 60 years of age and be a candidate for myeloablative donor stem cell transplantation
* Patients must receive myeloablative regimen using fludarabine and busulfan
* For related donors: The donor and recipient must have a 5/6 match at the HLA A, B, and DRB1 loci. [Patients with a 6/6 related donor are NOT eligible.] For unrelated donors: The donor and recipient must have a 5/6 or 6/6 match at the HLA A, B, and DRB1 loci.
* The typing level to define a match at the A and B locus must be at the level of mid-resolution DNA typing. The acceptable level to define a match at DRB1 will be by allelic typing by high resolution DNA sequencing.
* Any disease for which myeloablative transplantation is appropriate is eligible except: Progressive or poorly controlled malignancies for which the likelihood of durable disease control [i.e., patients expected to have at least 6 months PFS from date of transplant] is <25%.

Exclusion Criteria:

* Not a candidate for myeloablative conditioning regimen using the current BMT program clinical guidelines.
* Patient has a 6/6 HLA-matched related donor
* Karnofsky or Lansky performance status of < 60% at the time of admission for HSCT
* Patients with evidence of HIV infection or other opportunistic infection including but not limited to tuberculosis and histoplasmosis.
* Any conditions, in the opinion of the transplant team such as substance abuse, or severe personality disorder that would keep the patients from complying with the needs of the protocol and would markedly increase the morbidity and mortality from the procedure.
* Pregnancy.
* T-cell depleted allograft
* Patients with documented infections, not responding well to antibiotic therapy.
* Patients with bacteremia.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2004-08; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MD, MS, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Loyola University Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - The University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Background] Choi SW, Stiff P, Cooke K, Ferrara JL, Braun T, Kitko C, Reddy P, Yanik G, Mineishi S, Paczesny S, Hanauer D, Pawarode A, Peres E, Rodriguez T, Smith S, Levine JE. TNF-inhibition with etanercept for graft-versus-host disease prevention in high-risk HCT: lower TNFR1 levels correlate with better outcomes. Biol Blood Marrow Transplant. 2012 Oct;18(10):1525-32. doi: 10.1016/j.bbmt.2012.03.013. Epub 2012 Mar 30. PMID 22469883
- [Derived] Yanik GA, Mineishi S, Levine JE, Kitko CL, White ES, Vander Lugt MT, Harris AC, Braun T, Cooke KR. Soluble tumor necrosis factor receptor: enbrel (etanercept) for subacute pulmonary dysfunction following allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Jul;18(7):1044-54. doi: 10.1016/j.bbmt.2011.11.031. Epub 2011 Dec 10. PMID 22155140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted with recruitment taking place at the Blood and Marrow Transplantation Programs of the University of Michigan in Ann Arbor, Michigan and at Loyola University Medical Center, in Maywood, Illinois. The patients participating in this study, underwent transplantation, dating from April 2005-November 2009.
Pre-assignment Details: Patients >1 year of age who were candidates for a myeloablative allo-hemopoietic cell transplant were eligible for inclusion. Donors and recipients were required to match for 7/8 or 8/8 HLA-A, HLA-B, HLA-C, and HLA-DRB1 loci. Patients with an 8/8 HLA-matched related donor were not eligible.
Groups:
- GVHD Prophylaxis: GVHD prophylaxis with etanercept
  Etanercept : Etanercept 0.4 mg/kg per dose [maximum dose 25 mg] SC for prophylaxis. To start in the 24 hour time period along with the initiation of the preparative regimen for the stem cell transplant.
  Etanercept will be administered twice weekly until day +56 (8 weeks) post transplant.
Period: Overall Study
Arm/Group | GVHD Prophylaxis
Started | 100 (Number of evaluable patients)
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GVHD Prophylaxis
Number analyzed (Participants) | 100
Age, Continuous [Median (Full Range); unit: years] | 47 (5) [2 to 61]
Gender [Count of Participants; unit: Participants]
  Female | 43
  Male | 57
Region of Enrollment [Number; unit: participants]
  United States | 100
Disease status at transplantation [Number; unit: participants] — Disease classifications correspond to the Center for International Blood and Marrow Transplant Research Request for Information Disease Classifications Form (www.cibmtr.org).
  participants
    Low risk | 39
    Intermediate risk | 33
    High risk | 28
Donor match [Number; unit: participants]
  8/8 matched unrelated | 71
  7/8 mismatched unrelated | 26
  7/8 mismatched related | 3
Conditioning Regimen Parameter [Number; unit: participants] — Those subjects that did or did not receive Total body irradiation as part of their conditioning regimen.
  participants
    Non-Total body radiation | 71
    Total body radiation | 29

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Experiencing Acute GVHD After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Description: In order to determine whether etanercept, given prophylactically along with a standard Graft Versus Host Disease (GVHD) prevention regimen, will decrease the 100-day mortality and the rate of acute GVHD after allogeneic hematopoietic stem cell transplantation(HSCT), the incidence of grades 2-4 and grades 3-4 GVHD were calculated.
  GVHD can be clinically graded as 0, I, II, III, or IV. Definition of grades are:
  Grade 0 - No stage 1-4 of any organ Grade I - Stage 1-2 rash and no liver or gut involvement Grade II - Stage 3 rash, or Stage 1 liver involvement, or Stage 1 gastrointestinal involvement Grade III - Stage 0-3 skin, with STage 2-3 liver, or Stage 2-3 gastrointestinal involvement Grade IV - Stage 4 skin, liver, or gastrointestinal involvement
Time Frame: 100 days
Population: To provide Sufficient power
Measure: Number; unit: percentage of participants
Arm/Group | GVHD Prophylaxis
Number analyzed (Participants) | 100
percentage of participants
  Incidence of Grades 2-4 GVHD | 45 [95 to 105]
  Incidence of Grades 3-4 GVHD | 18

2. Secondary Outcome: Number of Patients Experiencing Etanercept Toxicity
Description: Toxicity of etanercept was evaluated by the following: the number of patients experiencing allergic reactions, the number of patients that discontinued etanercept early, the number of patients experiencing bacteremia, and the number of patients experiencing viral reactivations.
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | GVHD Prophylaxis
Number analyzed (Participants) | 100
participants
  Number of Patients Experiencing Allergic Reactions | 0
  Number of Patients that Discontinued Drug Early | 5
  Number of Patients Experiencing Bacteremia | 59
  Number of Patients Experiencing Viral Reactivation | 24

3. Secondary Outcome: The Number of Patients That Experience Idiopathic Pulmonary Syndrome (IPS)
Description: The Effect of etanercept on the incidence of idiopathic pulmonary syndrome (IPS). Patients who received Total Body Irradiation (TBI) transplant conditioning were compared to those who received another form of transplant conditioning.
Time Frame: 100 days
Population: TBI versus Non-TBI transplant conditioning
Measure: Count of Participants; unit: Participants
Groups:
- Total Body Irradiation (TBI): GVHD prophylaxis with etanercept in patients receiving Total Body Irradiation (TBI) transplant conditioning.
  Etanercept : Etanercept 0.4 mg/kg per dose [maximum dose 25 mg] SC for prophylaxis. To start in the 24 hour time period along with the initiation of the preparative regimen for the stem cell transplant.
  Etanercept will be administered twice weekly until day +56 (8 weeks) post transplant.
- Non-TBI: GVHD prophylaxis with etanercept
  Etanercept : Etanercept 0.4 mg/kg per dose [maximum dose 25 mg] SC for prophylaxis. To start in the 24 hour time period along with the initiation of the preparative regimen for the stem cell transplant.
  Etanercept will be administered twice weekly until day +56 (8 weeks) post transplant.
Arm/Group | Total Body Irradiation (TBI) | Non-TBI
Number analyzed (Participants) | 29 | 71
Participants | 1 | 0

4. Secondary Outcome: Day +7 TNFR1 Ratio in TBI-Treated Patients vs. Non-TBI-Treated Patients
Description: The effect of etanercept on plasma cytokine levels after Hematopoietic Stem Cell Transplantation (HSCT) was analyzed. Tumor Necrosis Factor Receptor 1 (TNFR1) ratios (TNFR1 posttransplantation day+7 / TNFR1pretransplantation baseline were calculated. Patients who received Total Body Irradiation (TBI) transplant conditioning were compared to those who received another form of transplant conditioning.
Time Frame: Day+7, post transplant
Population: TBI versus non-TBI transplant conditioning
Measure: Mean (Full Range); unit: TNFR1 Ratio
Arm/Group | Total Body Irradiation (TBI) | Non-TBI
Number analyzed (Participants) | 29 | 71
TNFR1 Ratio | 1.89 [1.07 to 5.15] | 1.1 [0.41 to 5.47]
Statistical Analysis 1: Comparison: Total Body Irradiation (TBI) vs Non-TBI; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Wilcoxon rank sum test

5. Secondary Outcome: The Impact of Tumor Necrosis Factor (TNF) Polymorphisms on Response to Therapy.
Time Frame: 100 days
Population: This was not analyzed in the population and there are no plans to analyze this in the future. The study is complete and the principal investigator has left the institution.
Arm/Group | Total Body Irradiation (TBI) | Non-TBI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the first dose of study drug until day +100 post transplant.
Arm/Group | GVHD Prophylaxis
Serious Adverse Events (participants affected / at risk) | 25/100
Other Adverse Events (participants affected / at risk) | 89/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVHD Prophylaxis (N=100)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic Reaction / Hypersensitivity (Immune system disorders) | 1 (1)
Blood Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2)
CNS Cerebrovascular Ischemia (Nervous system disorders) | 1 (2)
Catheter - Related Infection (Infections and infestations) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Infection wtih Unknown ANC (Infections and infestations) | 1 (1)
Infection without Neutropenia (Infections and infestations) | 6 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Personality / Behavioral (Psychiatric disorders) | 1 (1)
Rash / Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sexual / Reproductive Function (Reproductive system and breast disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Thrombosis / Embolism (Vascular disorders) | 1 (1)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVHD Prophylaxis (N=100)
Abdominal Pain or Cramping (Gastrointestinal disorders) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 24 (29)
Confusion (Psychiatric disorders) | 10 (12)
Constitutional Symptoms - Other (General disorders) | 7 (10)
Depressed Level of Consciousness (Nervous system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (17)
Edema (General disorders) | 11 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Fatigue (General disorders) | 14 (14)
Febrile Neutropenia (Blood and lymphatic system disorders) | 24 (24)
Hallucinations (Psychiatric disorders) | 10 (10)
Headache (Nervous system disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 30 (50)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (8)
Hypertension (Vascular disorders) | 24 (29)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (15)
Hypokalemia (Metabolism and nutrition disorders) | 18 (22)
Hyponatremia (Metabolism and nutrition disorders) | 11 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hypotension (Vascular disorders) | 22 (22)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 30 (35)
Infection with Grade 3 or 4 Neutropenia (Infections and infestations) | 11 (11)
Mood Alteration - Anxiety, Agitation (Psychiatric disorders) | 8 (9)
Mood Alteration - Depression (Psychiatric disorders) | 12 (12)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 9 (9)
Pain - Other (General disorders) | 5 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis / Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rash / Desquamation (Skin and subcutaneous tissue disorders) | 8 (8)
Renal Failure (Renal and urinary disorders) | 6 (6)
AST High (Investigations) | 6 (6)
ALT High (Investigations) | 11 (11)
Sinus Tachycardia (Cardiac disorders) | 8 (9)
Stomatitis Pharyngitis (Infections and infestations) | 18 (19)
Stomatitis Pharyngitis BMT (Infections and infestations) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No